CLINICAL TRIAL: NCT02982876
Title: Airway Stents for Excessive Dynamic Airway Collapse: A Randomized Controlled Trial
Brief Title: Airway Stents for Excessive Dynamic Airway Collapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Association of Broncology and Interventional Pulmonology (Unknown); Curetbm.org Fundation (Unknown); Hood Laboratories (Unknown); Boston Medical products inc (Unknown)
Responsible Party: Principal Investigator, Adnan Majid, MD, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000246
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2024-05

CONDITIONS: Tracheobronchomalacia; Excessive Dynamic Airway Collapse
Keywords: Silicone Airway stent; Metallic Airway stent
MeSH Terms: conditions — Tracheobronchomalacia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Management Group (No Intervention): The patients assigned to the medical management group will be placed on a scheduled institution protocol using mucolytic and expectorant therapy (nebulizer treatments using mucolytic (N-acetylcysteine) for 15 minutes BID, Guafenesin (Mucinex®) 1200 mg BID, codeine as needed and Flutter valve BID.
- Treatment group (Active Comparator): The patients assigned to treatment group will undergo flexible bronchoscopy with dynamic maneuvers, rigid bronchoscope , tracheobronchial wash and airway stent placement
  Interventions: Procedure: Dynamic Flexible Bronchoscopy; Procedure: Rigid Bronchoscopy; Device: Stent placement

INTERVENTIONS:
Procedure: Dynamic Flexible Bronchoscopy — The bronchoscope will be introduced into the proximal trachea at the level of the cricoid. At that point, patients will be instructed to take a deep breath, hold it and then blow it out (forced expiratory maneuver). Maneuvers will be done at the following six sites: proximal trachea at the level of the cricoid; mid-trachea 5 cm proximal to the carina; distal trachea 2 cm proximal to the carina; right main stem bronchus at the right tracheobronchial angle; bronchus intermedius and left main bronchus at the left tracheobronchial angle
  Arms: Treatment group
Procedure: Rigid Bronchoscopy — Under general anesthesia, a rigid bronchoscope (Bryan-Dumon Series II; Bryan Corporation; Woburn, MA) will be introduced, and respiration will be maintained through jet ventilation.
  Arms: Treatment group
Device: Stent placement — Silicone Y stent or uncovered self-expanding metallic stent will be placed in the standard fashion and good fit will be confirmed visually.
  Arms: Treatment group

SUMMARY:
Airway stents are used as standard of care to identify which patients with excessive dynamic airway collapse will benefit from a definitive surgical treatment. However, the specific way in which these stents are effective has not been tested. The purpose of this research study is to determine the effectiveness of airway stents when used in the airways of patients with severe symptomatic excessive dynamic airway collapse compared to patients with severe symptomatic excessive dynamic airway collapse that do not receive airway stent.

DETAILED DESCRIPTION:
Study Design

This randomized controlled trial will be conducted at Beth Israel Deaconess Medical Center (BIDMC) in accordance with Good Clinical Practice Standards and under IRB supervision. We plan to enroll total of 48 patients with EDAC randomized by a computer generated system to either intervention group (airway stent) or medical management group.

Description of the study

Previous to appointment all patients will have Airway CT scan, 6 minute walk test and pulmonary function test as per protocol and standard of care.

Enrollment

Patients with severe EDAC who remain symptomatic despite optimal medical management will be informed about the trial and if interested will be recruited for the study.

Operative Technique

Patients in the treatment group (stent) will undergo bronchoscopy under light sedation and rigid bronchoscopy under general anesthesia. The treatment group will undergo a bronchial wash and placement of an airway stent.Patients assigned to the medical management group will not undergo bronchoscopy.

Stents

Based on the patient's airway anatomy an uncovered self-expanding metallic stent (Ultraflex™ Single-Use Tracheobronchial Stent System) or a silicone Y-stent(Endoxane, Novatech S.A., Aubagne-France or Channick Hood Laboratories, Pembroke, MA, 02359) will be used in the study.

During Stent Trial

After bronchoscopy, patients in the treatment group will receive a standardized medication regimen to include mucolytics, cough suppressors and expectorants in order to decrease the risk of potential complications following the procedure.

Follow-up

All participants will be scheduled for a follow-up visit in the following 14 days either after rigid bronchoscopy (treatment group) or after first visit (medical management group) with 6MWTs and PFTs. In this visit all patients will be asked to complete the SGRQ, CQLQ and mMRC questionnaires by the research team. All this data will be recorded in an encrypted database. Afterwards, the patients in the medical management arm will be offered a stent trial as part of standard of care.

Stent removal

The patients from the treatment arm will be scheduled for a rigid bronchoscopy, stent removal and bronchial lavage under anesthesia in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Patient with sever symptomatic EDAC (collapse >90% of the airway during exhalation at dynamic CT scan)
* Age > 18 years

Exclusion Criteria:

* Patients who have not been well managed from their respiratory comorbidities (asthma, COPD, obstructed sleep apnea, GERD, relapsing polychondritis)
* Current respiratory infection
* Resting bradycardia (<50 beats/min), frequent multifocal PVCs, complex ventricular arrhythmia, sustained SVT
* Dysrhythmia that might pose a risk during exercise or training
* Any disease or condition that interferes with completion of initial or follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire | 7-14 days
  Index designed to measure health status in patients with respiratory symptoms

SECONDARY OUTCOMES:
modified Medical Research Council scale of dyspnea | 7-14 days
  Shortness of breath scale
Cough Quality of life Questionnaire | 7-14 days
6 minute walk test | 7-14 days
FEV1 | 7-14 days
Peak flow | 7-14 days
Self-reported symptoms | 7-14 days
  dyspnea, inability to clear secretions, cough, recurrent infection and wheezing.
Complications | 7-14 days
  Airway infections

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Majid, MD, Principal Investigator — Beth Israel Deaconess Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leong P, Bardin PG, Lau KK. What's in a name? Expiratory tracheal narrowing in adults explained. Clin Radiol. 2013 Dec;68(12):1268-75. doi: 10.1016/j.crad.2013.06.017. Epub 2013 Aug 13. PMID 23953005
- [Background] Murgu S, Colt H. Tracheobronchomalacia and excessive dynamic airway collapse. Clin Chest Med. 2013 Sep;34(3):527-55. doi: 10.1016/j.ccm.2013.05.003. Epub 2013 Jun 27. PMID 23993822
- [Background] Ridge CA, O'donnell CR, Lee EY, Majid A, Boiselle PM. Tracheobronchomalacia: current concepts and controversies. J Thorac Imaging. 2011 Nov;26(4):278-89. doi: 10.1097/RTI.0b013e3182203342. PMID 22009081
- [Background] Boiselle PM, O'Donnell CR, Bankier AA, Ernst A, Millet ME, Potemkin A, Loring SH. Tracheal collapsibility in healthy volunteers during forced expiration: assessment with multidetector CT. Radiology. 2009 Jul;252(1):255-62. doi: 10.1148/radiol.2521081958. Epub 2009 May 6. PMID 19420322
- [Background] Carden KA, Boiselle PM, Waltz DA, Ernst A. Tracheomalacia and tracheobronchomalacia in children and adults: an in-depth review. Chest. 2005 Mar;127(3):984-1005. doi: 10.1378/chest.127.3.984. PMID 15764786
- [Background] Jokinen K, Palva T, Nuutinen J. Chronic bronchitis. A bronchologic evaluation. ORL J Otorhinolaryngol Relat Spec. 1976;38(3):178-86. doi: 10.1159/000275273. PMID 945891
- [Background] Palombini BC, Villanova CA, Araujo E, Gastal OL, Alt DC, Stolz DP, Palombini CO. A pathogenic triad in chronic cough: asthma, postnasal drip syndrome, and gastroesophageal reflux disease. Chest. 1999 Aug;116(2):279-84. doi: 10.1378/chest.116.2.279. PMID 10453852
- [Background] Ikeda S, Hanawa T, Konishi T, Adachi M, Sawai S, Chiba W, Kosaba S, Hatakenaka R, Matsubara Y, Funatsu T. [Diagnosis, incidence, clinicopathology and surgical treatment of acquired tracheobronchomalacia]. Nihon Kyobu Shikkan Gakkai Zasshi. 1992 Jun;30(6):1028-35. Japanese. PMID 1507676
- [Background] Majid A, Gaurav K, Sanchez JM, Berger RL, Folch E, Fernandez-Bussy S, Ernst A, Gangadharan SP. Evaluation of tracheobronchomalacia by dynamic flexible bronchoscopy. A pilot study. Ann Am Thorac Soc. 2014 Jul;11(6):951-5. doi: 10.1513/AnnalsATS.201312-435BC. PMID 24960030
- [Background] Lee KS, Sun MRM, Ernst A, Feller-Kopman D, Majid A, Boiselle PM. Comparison of Dynamic Expiratory CT With Bronchoscopy for Diagnosing Airway Malacia: A Pilot Evaluation. Chest. 2007 Mar;131(3):758-764. doi: 10.1378/chest.06-2164. PMID 17356090
- [Background] Ernst A, Majid A, Feller-Kopman D, Guerrero J, Boiselle P, Loring SH, O'Donnell C, Decamp M, Herth FJ, Gangadharan S, Ashiku S. Airway stabilization with silicone stents for treating adult tracheobronchomalacia: a prospective observational study. Chest. 2007 Aug;132(2):609-16. doi: 10.1378/chest.06-2708. PMID 17699133
- [Background] Litmanovich D, O'Donnell CR, Bankier AA, Ernst A, Millett ME, Loring SH, Boiselle PM. Bronchial collapsibility at forced expiration in healthy volunteers: assessment with multidetector CT. Radiology. 2010 Nov;257(2):560-7. doi: 10.1148/radiol.10100219. Epub 2010 Sep 9. PMID 20829540
- [Background] Majid A, Sosa AF, Ernst A, Feller-Kopman D, Folch E, Singh AK, Gangadharan S. Pulmonary function and flow-volume loop patterns in patients with tracheobronchomalacia. Respir Care. 2013 Sep;58(9):1521-6. doi: 10.4187/respcare.02277. Epub 2013 Mar 12. PMID 23481440
- [Background] Tamura Y, Sakatani K, Yamakoshi N, Terada H, Honda H, Komori C, Kuhara H, Morishita N, Shishido K, Matsuoka H, Shishido N, Ishihara H. [A case of severe COPD associated with tracheo-bronchial stenosis, treated with non-invasive positive pressure ventilation]. Nihon Kokyuki Gakkai Zasshi. 2008 Nov;46(11):915-20. Japanese. PMID 19068766
- [Background] Ferguson GT, Benoist J. Nasal continuous positive airway pressure in the treatment of tracheobronchomalacia. Am Rev Respir Dis. 1993 Feb;147(2):457-61. doi: 10.1164/ajrccm/147.2.457. PMID 8430971
- [Background] Adliff M, Ngato D, Keshavjee S, Brenaman S, Granton JT. Treatment of diffuse tracheomalacia secondary to relapsing polychondritis with continuous positive airway pressure. Chest. 1997 Dec;112(6):1701-4. doi: 10.1378/chest.112.6.1701. PMID 9404780
- [Background] Wright CD. Tracheomalacia. Chest Surg Clin N Am. 2003 May;13(2):349-57, viii. doi: 10.1016/s1052-3359(03)00036-x. PMID 12755319
- [Background] Gangadharan SP, Bakhos CT, Majid A, Kent MS, Michaud G, Ernst A, Ashiku SK, DeCamp MM. Technical aspects and outcomes of tracheobronchoplasty for severe tracheobronchomalacia. Ann Thorac Surg. 2011 May;91(5):1574-80; discussion 1580-1. doi: 10.1016/j.athoracsur.2011.01.009. Epub 2011 Mar 5. PMID 21377650
- [Background] Majid A, Guerrero J, Gangadharan S, Feller-Kopman D, Boiselle P, DeCamp M, Ashiku S, Michaud G, Herth F, Ernst A. Tracheobronchoplasty for severe tracheobronchomalacia: a prospective outcome analysis. Chest. 2008 Oct;134(4):801-807. doi: 10.1378/chest.08-0728. PMID 18842912
- [Background] Ernst A, Odell DD, Michaud G, Majid A, Herth FFJ, Gangadharan SP. Central airway stabilization for tracheobronchomalacia improves quality of life in patients with COPD. Chest. 2011 Nov;140(5):1162-1168. doi: 10.1378/chest.10-3051. Epub 2011 Aug 25. PMID 21868463
- [Background] Murgu SD, Colt HG. Complications of silicone stent insertion in patients with expiratory central airway collapse. Ann Thorac Surg. 2007 Dec;84(6):1870-7. doi: 10.1016/j.athoracsur.2007.07.026. PMID 18036901
- [Background] Machuzak M, Santacruz JF, Gildea T, Murthy SC. Airway complications after lung transplantation. Thorac Surg Clin. 2015;25(1):55-75. doi: 10.1016/j.thorsurg.2014.09.008. PMID 25430430
- [Background] Chhajed PN, Malouf MA, Tamm M, Spratt P, Glanville AR. Interventional bronchoscopy for the management of airway complications following lung transplantation. Chest. 2001 Dec;120(6):1894-9. doi: 10.1378/chest.120.6.1894. PMID 11742919
- [Background] Zhang J, Hasegawa I, Feller-Kopman D, Boiselle PM. 2003 AUR Memorial Award. Dynamic expiratory volumetric CT imaging of the central airways: comparison of standard-dose and low-dose techniques. Acad Radiol. 2003 Jul;10(7):719-24. doi: 10.1016/s1076-6332(03)80117-4. PMID 12862281
- [Background] Odell DD, Majid A, Gangadharan SP, Ernst A. Adoption of a standardized protocol decreases serious complications of airway stenting in patients with tracheobronchomalacia. Chest. 2010; 138(suppl 4):A784
- [Background] Jones PW, Quirk FH, Baveystock CM. The St George's Respiratory Questionnaire. Respir Med. 1991 Sep;85 Suppl B:25-31; discussion 33-7. doi: 10.1016/s0954-6111(06)80166-6. PMID 1759018
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Background] French CT, Irwin RS, Fletcher KE, Adams TM. Evaluation of a cough-specific quality-of-life questionnaire. Chest. 2002 Apr;121(4):1123-31. doi: 10.1378/chest.121.4.1123. PMID 11948042
- [Background] Jones PW. St. George's Respiratory Questionnaire: MCID. COPD. 2005 Mar;2(1):75-9. doi: 10.1081/copd-200050513. PMID 17136966
- [Background] Donohue JF. Minimal clinically important differences in COPD lung function. COPD. 2005 Mar;2(1):111-24. doi: 10.1081/copd-200053377. PMID 17136971
- [Background] Puhan MA, Chandra D, Mosenifar Z, Ries A, Make B, Hansel NN, Wise RA, Sciurba F; National Emphysema Treatment Trial (NETT) Research Group. The minimal important difference of exercise tests in severe COPD. Eur Respir J. 2011 Apr;37(4):784-90. doi: 10.1183/09031936.00063810. Epub 2010 Aug 6. PMID 20693247
- [Background] de Torres JP, Pinto-Plata V, Ingenito E, Bagley P, Gray A, Berger R, Celli B. Power of outcome measurements to detect clinically significant changes in pulmonary rehabilitation of patients with COPD. Chest. 2002 Apr;121(4):1092-8. doi: 10.1378/chest.121.4.1092. PMID 11948037
- [Background] Fletcher KE, French CT, Irwin RS, Corapi KM, Norman GR. A prospective global measure, the Punum Ladder, provides more valid assessments of quality of life than a retrospective transition measure. J Clin Epidemiol. 2010 Oct;63(10):1123-31. doi: 10.1016/j.jclinepi.2009.09.015. Epub 2010 Mar 19. PMID 20303709
- [Background] Nouraei SM, Franco RA, Dowdall JR, Nouraei SA, Mills H, Virk JS, Sandhu GS, Polkey M. Physiology-based minimum clinically important difference thresholds in adult laryngotracheal stenosis. Laryngoscope. 2014 Oct;124(10):2313-20. doi: 10.1002/lary.24641. Epub 2014 Apr 4. PMID 25265276
- [Background] Shlomi D, Peled N, Shitrit D, Bendayan D, Amital A, Kramer MR. Protective effect of immunosuppression on granulation tissue formation in metallic airway stents. Laryngoscope. 2008 Aug;118(8):1383-8. doi: 10.1097/MLG.0b013e318172d686. PMID 18496158
- [Background] Jones PW. Interpreting thresholds for a clinically significant change in health status in asthma and COPD. Eur Respir J. 2002 Mar;19(3):398-404. doi: 10.1183/09031936.02.00063702. PMID 11936514